CLINICAL TRIAL: NCT06538077
Title: Branch Chain Amino Acids vs. Rifaximin in Patients With Cirrhosis for Secondary Prophylaxis of Hepatic Encephalopathy: Double-blind Placebo-controlled Multicentric Randomized Controlled Trial
Brief Title: BCAA vs. Rifaximin in Patients With Cirrhosis for Secondary Prophylaxis of HE
Acronym: HERB
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Principal Investigator, Madhumita Premkumar, ASSOCIATE PROFESSOR, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PGI/HEP/567
Record Dates: First submitted 2024-04-23; First posted 2024-08-05 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Hepatic Encephalopathy; Decompensated Cirrhosis; Minimal Hepatic Encephalopathy
Keywords: Hepatic encephalopathy; Branched-chain amino acids; Computerized neurocognitive test battery; Double blind placebo controlled multicentric randomized controlled trial; rifaximin
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Amino Acids, Branched-Chain; Rifaximin; Lactulose

STUDY DESIGN:
Intervention Model Description: In addition to the BCAA vs Rifaximin, both groups will be treated with 30-60 ml lactulose three times a day to ensure passage of 2-3 semisoft stools per day.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind double dummy placebo-controlled multicentric randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A1=Experimental: (Experimental): Drug: Oral BCAA + Rifaximin placebo + Lactulose ( Oral BCAA 15 gm in once daily dose With Lactulose for 12 weeks)
  Interventions: Drug: Oral Branched chain Amino acid; Drug: Lactulose; Drug: Placebo for Rifaximin 550mg
- A2= Experimental: (Experimental): Drug: Rifaximin+ BCAA Placebo + Lactulose ( Oral Rifaximin 550 mg twice daily daily + Lactulose therapy for 12 weeks)
  Interventions: Drug: Rifaximin 550 MG; Drug: Lactulose; Drug: Placebo for BCAA

INTERVENTIONS:
Drug: Oral Branched chain Amino acid — The active drug BCAA supplement will be dispensed in a dose of 15 gm once daily x 12 weeks
  Arms: A1=Experimental:
Drug: Rifaximin 550 MG — Active drug rifaximin will be dispensed in a dose of 550mg twice daily x 12 weeks
  Arms: A2= Experimental:
Drug: Lactulose — Both groups will be treated with will be treated with 30-60 ml lactulose three times a day to ensure passage of 2-3 semisoft stools per day
Drug: Placebo for BCAA — A placebo comparator of 15 gm of skimmed milk powder will be used.
  Arms: A2= Experimental:
Drug: Placebo for Rifaximin 550mg — Identical placebo sugar pills will be used as a placebo.
  Arms: A1=Experimental:

SUMMARY:
Rationale

* Patients who recover from an episode of overt HE(OHE) are at risk of recurrent episodes of HE and persistent minimal hepatic encephalopathy, impacting their daily functioning and mental health.
* A multicentric pan-India team will evaluate the role of oral branched-chain amino acids (BCAA) vs Rifaximin as secondary prophylaxis following overt HE as compared with improvement in cognitive function.

Novelty:

* This study is intended to investigate the role of BCAA vs rifaximin as the ideal second-line therapy for HE management, recurrence, and overall health, including cognitive function, depression and anxiety.
* The head-to-head comparison of BCAA+lactulose+ pill-placebo vs rifaximin+ lactulose+ powder-placebo ensures minimization of bias and has adequate power to determine rates of recurrence,

Objectives:

* To assess the 1st breakthrough episode of HE during 6months in BCAA vs rifaximin groups as ideal secondary prophylaxis in HE. Methodology
* Double-blind placebo-controlled double-dummy randomized trial of BCAA supplementation vs rifaximin as the ideal second-line therapy in patients with cirrhosis who have recovered from an episode of OHE. Expected Outcome
* Ideal second line agent HE prophylaxis (rifaximin or BCAA) following 1st line lactulose is unclear in an Indian context where dysbiosis and sarcopenia are prevalent, and cost of therapy needs to be optimized.
* Optimal HE management prevents recurrence episodes of HE, and improves prognosis, neurocognitive function, and overall health-related quality of life(HRQOL).
* Creation of a management algorithm based deductive models incorporating etiology and severity of liver disease, cognitive performance, sarcopenia, and ammonia, and neuropsychiatric impact of using BCAA vs Rifaximin will be created.

DETAILED DESCRIPTION:
Hepatic encephalopathy (HE), a complex neuropsychiatric syndrome arising from liver dysfunction and the establishment of portosystemic shunts (PSS), presents a significant clinical challenge, marked by a spectrum of cognitive, emotional, and motor disturbances. These conditions necessitate precise diagnostic and therapeutic approaches to mitigate its impact on patient well-being and quality of life.

* The prevalence of OHE at the time of diagnosis of cirrhosis is 10%-14% in general, 16%-21% in those with decompensated cirrhosis. The cumulated numbers indicate that OHE will occur in 30%-40% of those with cirrhosis at some time during their clinical course and in the survivors in most cases repeatedly. Minimal HE (MHE) or covert HE (CHE) occurs in 20%-80% of patients with cirrhosis. This high incidence rate calls for effective, accessible, and cost-efficient treatment modalities to improve patient outcomes and quality of life.
* Indian patients have sarcopenia and reduced muscle strength impairing peripheral ammonia metabolism, and also have gut dysbiosis which can predispose to another episode of HE. A critical initial step in addressing HE involves the identification of precipitating factors, with evidence suggesting that reversible elements contribute to over 80% of HE cases.
* Current therapeutic interventions primarily target the reduction of blood ammonia levels, yet the effectiveness of these treatments varies, underscoring the necessity for ongoing research and innovation in HE management.
* Patients recovering from OHE are at risk of recurrent episodes and may suffer from persistent MHE, a condition often undiagnosed due to its subtle cognitive manifestations. Such individuals may have cognitive impairment that affect patients' daily functioning and mental health, necessitating the development of standardized diagnostic psychometric tests protocols tailored to diverse populations.
* Mainstay for treatment of HE has been lactulose or lactitol. How lactulose acts in HE has been a matter of debate and various hypotheses have been postulated. Inglefenger et al., suggested it to be due to proliferation of Lactobacillus with inhibition of Bacteroides and other organisms (28). Lactulose has pleiotropic effects, and reduction of ammonia is only one of the ways in which it acts on HE.
* Rifaximin is an oral antibiotic having <0.4% of systemic absorption. It acts against coliforms like Escherichia coli and plays a role in the reduction of ammonia levels and prevention of recurrence of HE . Several trials have compared Rifaximin as a therapy of HE with placebo, neomycin and non-absorbable disaccharides . Rifaximin emerged as a promising alternative, showing comparable efficacy in managing OHE and preventing its recurrence..
* This is a double-blind, randomized placebo-controlled trial of branched-chain amino acid supplementation vs rifaximin as the ideal second-line therapy in patients with cirrhosis who have recovered from an episode of overt hepatic encephalopathy, with either drug given over 12 weeks with endpoints being prevention of recurrence of another episode of HE, efficacy, safety, and improvement in neurocognitive function

ELIGIBILITY:
Inclusion Criteria:

1. Cirrhosis defined by standard clinical, ultrasonographic findings and/or histological criteria. Cirrhosis of any etiology may be included. However, patients with cirrhosis due to autoimmune hepatitis must be on stable corticosteroid doses for ≥3-month period before study inclusion; those with viral hepatitis, must similarly be on anti-viral therapy with controlled viremia or with SVR.
2. Any gender
3. Discharged from the hospital following an episode of overt hepatic encephalopathy.
4. Participants able to give informed consent

Exclusion Criteria:

1. Subjects with active bacterial or fungal infection
2. Subjects with active or very recent gastrointestinal bleeding in the last 2 weeks.
3. Current overt hepatic encephalopathy, defined as grade II-IV hepatic encephalopathy according to the West-Haven classification.
4. Conditions that can impact interpretation of cognitive function:

   i) Untreated viremic hepatitis C virus infection ii) Established neurological/degenerative disorders iii) Patient undergoing active alcohol withdrawal treatment Iv) Patient is intoxicated or under the influence of illicit drugs as per clinician assessment V) Treatment with antipsychotics or other psychotropic drugs with sedative effects
5. Patients with active hepatocellular carcinoma or history of hepatocellular carcinoma that is in remission for less than six months.
6. Patients with a history of significant extrahepatic disease with impaired short-term prognosis, including: i) Congestive heart failure New York Heart Association Grade III/IV or ejection fraction<30% ii) COPD: GOLD >2, ii) Chronic kidney disease with serum creatinine >2mg/dL or under renal replacement therapy.
7. Patients with current extra hepatic malignancies, including solid tumours and hematologic disorders.
8. Patients with MELD>20
9. Patients with mental incapacity, or those unlikely to survive 12 weeks or any other reason considered by the investigator precluding adequate understanding, cooperation, or compliance in the study activities.
10. Patients with TIPS shunt in situ
11. Pregnancy (urine pregnancy test at inclusion)
12. Refusal or inability to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Number of breakthrough event of overt hepatic encephalopathy in BCAA vs rifaximin arm | 24 Weeks
  Time to a breakthrough overt HE episode will be the duration (number of days) from time of first dose of study drug to the first breakthrough overt HE episode. The number of events of a first breakthrough overt HE episode during the treatment period will be assessed

SECONDARY OUTCOMES:
Computerized Cognitive Test battery for Cognitive performance | At Enrolment
  A curated Computer based Cognitive test battery has been created for this protocol with a fixed set of tasks comprising Animal Naming Test, reaction times, digit span and number connection tests. This has been designed using the PEBL opensource language. Psychology Experiment Building Language. [2019-03] PEBL Version 2.1. The battery has been validated by us previously in patients with chronic hepatitis C infection.
Computerized Cognitive Test battery for Cognitive performance | 30 days
  Computerized Cognitive Test battery: A curated Computer based Cognitive test battery has been created for this protocol with a fixed set of tasks comprising Animal Naming Test, reaction times, digit span and number connection tests. This has been designed using the PEBL opensource language. Psychology Experiment Building Language. [2019-03] PEBL Version 2.1. The battery has been validated by us previously in patients with chronic hepatitis C infection.
Computerized Cognitive Test battery for Cognitive performance | 90 days
  Computerized Cognitive Test battery A curated Computer based Cognitive test battery has been created for this protocol with a fixed set of tasks comprising Animal Naming Test, reaction times, digit span and number connection tests. This has been designed using the PEBL opensource language. Psychology Experiment Building Language. [2019-03] PEBL Version 2.1. The battery has been validated by us previously in patients with chronic hepatitis C infection.
Psychiatric Assessment | 0 days
  Beck's Depression Inventory (BDI) test will be performed. The scoring is as follows 1-10: These ups and downs are considered normal 11-16: Mild mood disturbance 17-20: Borderline clinical depression 21-30: Moderate depression31-40: Severe depression 40: Extreme depression
Psychiatric Assessment | 0 days
  Generalized anxiety disorder (GAD 7 score) will be performed. It has 7 questions. Using the threshold score of 10, the GAD-7 has a sensitivity of 89% and a specificity of 82% for GAD
Psychiatric Assessment | 30 days
  Generalized anxiety disorder (GAD 7 score) test will be performed
Psychiatric Assessment | 30 days
  Beck's Depression Inventory (BDI) test will be performed. The scoring is as follows 1-10: These ups and downs are considered normal 11-16: Mild mood disturbance 17-20: Borderline clinical depression 21-30: Moderate depression31-40: Severe depression 40: Extreme depression
Psychiatric Assessment | 90 days
  Beck's Depression Inventory (BDI)test will be performed The scoring is as follows 1-10: These ups and downs are considered normal 11-16: Mild mood disturbance 17-20: Borderline clinical depression 21-30: Moderate depression31-40: Severe depression 40: Extreme depression
Psychiatric Assessment | 90 days
  Generalized anxiety disorder (GAD 7 score) tests will be performed
HRQOL will be performed by SF-36 | 0 days
  Health related query of life will be performed.
HRQOL will be performed by SF-36 | 30 days
  Health related query of life will be performed.
HRQOL will be performed by SF-36 | 90 days
  Health related query of life will be performed.
Assessment of changes in ammonia | At enrolment
  Estimation of ammonia by arterial fasting test/ capillary test will be performed
Assessment of changes in ammonia | 24 week
  Estimation of ammonia by arterial fasting test/ capillary test will be performed
Assessment of changes in muscle health | Baseline
  Estimation of sarcopenia will be performed by muscle ultrasound by SARCUS.
Assessment of changes in muscle health | 30 days
  Estimation of sarcopenia by muscle ultrasound by SARCUS.
Assessment of changes in muscle health | 90 days
  Estimation of sarcopenia by muscle ultrasound by SARCUS.

CONTACTS AND LOCATIONS:
Locations (1):
- PGIMER, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No